CLINICAL TRIAL: NCT05571202
Title: Pain Score and Urine Retention Rate Between Spinal and General Anesthesia for Anorectal Surgery, Retrospective Observation Study
Brief Title: Urine Retention Rate Between Spinal and General Anesthesia for Anorectal Surgery
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CG22204A
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Anorectal Disorder
Keywords: anorectal surgery, hemorrhoid, anesthesia
MeSH Terms: conditions — Rectal Diseases; Hemorrhoids | interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Anorectal surgery patient under general anesthesia plus local infiltration: Anorectal surgery patient under general anesthesia plus local infiltration
  Interventions: Procedure: General anesthesia plus local infiltration
- Anorectal surgery patient under spinal anesthesia: Anorectal surgery patient under spinal anesthesia alone
  Interventions: Procedure: Spinal anesthesia

INTERVENTIONS:
Procedure: General anesthesia plus local infiltration — The eligible patients underwent anorectal surgery under general anesthesia (GE, GM, IVG) plus locally injected analgesics.
  Groups: Anorectal surgery patient under general anesthesia plus local infiltration
Procedure: Spinal anesthesia — The eligible patients underwent anorectal surgery under spinal anesthesia alone.
  Groups: Anorectal surgery patient under spinal anesthesia

SUMMARY:
Anorectal surgery includes pilonidal sinus, hemorrhoidectomy, anal fissure, and anal fistula operations. General and spinal anesthesia were common anesthetic methods in anorectal surgery. We designed this study to test the hypothesis that general anesthesia was superior than spinal anesthesia with respect to urine retention rate, pain score, recovery time, and side effects.

DETAILED DESCRIPTION:
Anorectal surgery includes pilonidal sinus, hemorrhoidectomy, anal fissure, and anal fistula operations. Deep level of anesthesia is required for these surgeries. Excellent operation conditions and rapid recovery is anticipated for optimal anesthesia. Various surgical and anesthetic techniques, including spinal anesthesia, general anesthesia and local infiltration have been used to increase the level of patients' perioperative analgesia and decrease the length of stay in the hospital. Among them, general and spinal anesthesia were common anesthetic methods in anorectal surgery. We designed this study to test the hypothesis that general anesthesia was superior than spinal anesthesia with respect to urine retention rate, pain score, recovery time, and side effects.

Inclusion Criteria:

* >20 years old patients
* ASA 1-2 patients
* Patients who will undergo anorectal surgery with including hemorrhoidectomy, fistulectomy, fistulotomy, fissurectomy and anoplasty.

Exclusion Criteria:

* Having known hypersensitivity to amide type local anesthetics
* Patients ASA >=3
* Surgery methods: hemorrhoidopexy, Laser hemorrhoidoplasty
* Fournier gangrene patients
* Surgery due to previous complications.

Characteristic data

1. Age, Gender, ASA class,
2. Past history: medical history, surgical history
3. Previous anorectal history
4. Type of anorectal surgery, number of hemorrhoidectomy
5. Methods of anesthesia, posture during surgery
6. Postoperative recovery room record: vital sign, Post Anaesthetic Discharge Scoring System (0-10, >9 can discharge)
7. Ward record: vital sign and urine retention need foley catherization

ELIGIBILITY:
Inclusion Criteria:

* >20 years old patients
* ASA 1-2 patients
* Patients who will undergo anorectal surgery with including hemorrhoidectomy, fistulectomy, fistulotomy, fissurectomy and anoplasty.

Exclusion Criteria:

* Having known hypersensitivity to amide type local anesthetics
* Patients ASA >=3
* Surgery methods: hemorrhoidopexy, Laser hemorrhoidoplasty
* Fournier gangrene patients
* Surgery due to previous complications

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Benign anorectal disease patients underwent surgery interventions. Characteristics of age, gender, height, weight, ASA score, past medical history, operational history were recorded from EHIS systems. Intraoperative findings which include anesthesia time, operation time, intraoperative fluid. Surgical outcomes include surgery complications, anesthesia complications, pain score. All of above data were retrospective recorded from hospital discharge note, OPD records, operation note, pathology report.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Urine retention rate | 0-24 hours post operation.
  urine retention events needs foley catheterization
Pain score | 0-24 hours post operation.
  Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
surgery complications | 0-30 days post operative days.
  surgery complications
anesthesia complications | 0-30 days post operative days.
  anesthesia complications rate

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Lin, M.D., Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Verterans General Hospital, Taichung, Taiwan